CLINICAL TRIAL: NCT04215133
Title: Inspiratory Muscle Training Versus Calf Muscle on Venous Function in Patients With Chronic Venous Insufficiency
Brief Title: Inspiratory Muscle Training Versus Calf Muscle on Venous Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gamze Aydin, Principal İnvestigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUCe
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Venous Insufficiency
Keywords: venous insufficiency; exercise therapy; inspiratory muscle; kalf muscle; venous return
MeSH Terms: conditions — Venous Insufficiency | interventions — Exercise Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- İnspiratory muscle training group (Experimental)
  Interventions: Other: exercise therapy
- Calf muscle training group (Experimental)
  Interventions: Other: exercise therapy
- Control (No Intervention)

INTERVENTIONS:
Other: exercise therapy — inspiratory muscle training consists of strengthening exercise with threshold Inspiratory muscle training device and calf muscle training consist of isotonic and isometric strengthening exercise for calf muscle. All groups will receive compression therapy at the same time.
  Arms: Calf muscle training group; İnspiratory muscle training group

SUMMARY:
The aim of this study was to evaluate the effect of exercise training in addition to compression therapy on quality of life, venous return time, muscle strength, clinical severity, functional capacity in venous insufficiency compared to compression treatment alone. Fourty-two volunteer patients with venous insufficiency will include in the study were randomly divided into three groups as inspiratory exercise, calf muscle exercise and control. While the control group will receive only compression therapy, the inspiratory exercise group will apply inspiratory muscle training consisted of strengthening exercise in addition to compression therapy; kalf muscle exercise group will apply strengthening exercise for calf muscle in addition to compression therapy for 2 days/week with physiotherapist and 3 days/week by themselves, 8 weeks. All the patients will assess with Chronic Venous Disease Quality of life Questionnaire-20 (CIVIQ-20), Nottingham Health Profile, Photopletismograph, Venous Clinical Severity Score (VCSS), hand-held dynamometer, Visual Analogue Scale (VAS), circumference measurements, 6-minute walk test (6MWT), before and after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of venous insufficiency between 18-75 years with duplex ultrasound imaging
* CEAP classification used in venous insufficiency is C2-C3-C4-C5
* Having written and verbal communication in Turkish

Exclusion Criteria:

* Acute deep vein thrombosis
* The presence of ulceration
* Being in class III and IV according to the New York Heart Association classification
* Presence of respiratory failure
* Undergoing chemotherapy due to the presence of any cancer
* Being in the process of treatment for neurological, orthopedic or rheumatologic diseases including lower extremity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-20 (Estimated)

PRIMARY OUTCOMES:
The Chronic Venous Insufficiency Questionnaire-20 (CIVIQ-20) | 12 months
  Quality of life
Photoplethysmograph (PPG) | 12 months
  venous return time

SECONDARY OUTCOMES:
Hand held dynamometer | 12 months
  muscle strength
Venous Clinical Severity Score (VCSS) | 12 months
  clinical severity
6 minutes walk test | 12 months
  functional capacity
digital goniometer | 12 months
  range of motion of ankle
visual analog scale | 12 months
  pain

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aydin G, Yeldan I, Akgul A, Ipek G. Effects of inspiratory muscle training versus calf muscle training on quality of life, pain, venous function and activity in patients with chronic venous insufficiency. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1137-1146. doi: 10.1016/j.jvsv.2022.04.012. Epub 2022 Jun 14. PMID 35710091